CLINICAL TRIAL: NCT04248426
Title: A Phase 1 Double-Blinded Study for Safety, Tolerability, Pharmacokinetics, and Antiviral Activity of ATI-2173 in Healthy Subjects and Subjects With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Antios Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANTT101
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATI-2173 (Experimental)
  Interventions: Drug: ATI-2173
- ATI-2173 Placebo (Placebo Comparator)
  Interventions: Drug: ATI-2173 Placebo

INTERVENTIONS:
Drug: ATI-2173 — ATI-2173 is a liver-targeted phosphoramidate prodrug of clevudine designed to enhance anti-HBV activity while decreasing systemic exposure to clevudine. It will be dosed as a capsule by mouth.
  Arms: ATI-2173
Drug: ATI-2173 Placebo — ATI-2173 Placebo is used as an inactive comparator to ATI-2173. It will be dosed as a capsule by mouth.
  Arms: ATI-2173 Placebo

SUMMARY:
This is a double-blinded, randomized, placebo-controlled study of safety, tolerability, pharmacokinetics, and antiviral activity in both healthy volunteers and volunteers with chronic hepatitis B virus infection. Healthy volunteers will be administered either a single oral dose or multiple oral doses of ATI-2173 and assessed for safety and tolerability including blood tests to show how the body metabolizes and eliminates the investigational drug. Volunteers with a diagnosis of chronic hepatitis B virus infection will be administered multiple oral doses of ATI-2173 and assessed for safety and tolerability including blood tests to show how the body metabolizes and eliminates the investigational drug as well as how the drug effects the virus infection.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Provision of signed and dated informed consent form (ICF)
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. If female, meets 1 of the following criteria:

   1. Is of childbearing potential and agrees to use an accepted contraceptive method. Acceptable method of contraception include:

      * Abstinence from heterosexual intercourse from at least 28 days prior to the first study drug administration through to at least 30 days after the last dose of the study drug or until completion of the study, whichever is longer
      * Male partner vasectomized at least 6 months prior to the first study drug administration
      * Use a systemic contraceptive or an intrauterine device (with or without hormones), from at least 28 days prior to the first study drug administration through to at least 30 days after the last dose of the study drug or until completion of the study, whichever is longer, with a male condom or a diaphragm/cervical cap plus spermicide, from the first study drug administration through to at least 30 days after the last dose of the study drug or until completion of the study, whichever is longer Or
   2. Male partner has had a vasectomy less than 6 months prior to dosing, and agrees to use an additional acceptable contraceptive method from the first study drug administration through to at least 30 days after the last dose of the study drug or until completion of the study, whichever is longer Or
   3. Is of non-childbearing potential, defined as surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (i.e. at least 1 year without menses without an alternative medical condition prior to the first study drug administration and follicle-stimulating hormone levels ≥ 40 mIU/mL at screening)
4. If male, meets 1 of the following criteria:

   1. Is able to procreate and agrees to use 1 of the accepted contraceptive regimens and not to donate sperm from the first study drug administration to at least 90 days after the last drug administration. An acceptable method of contraception includes 1 of the following:

      * Abstinence from heterosexual intercourse
      * Male condom with spermicide or male condom with a vaginal spermicide (gel, foam, or suppository) or
   2. Is unable to procreate; defined as surgically sterile (i.e. has undergone a vasectomy at least 180 days prior to the first study drug administration)
5. Light-, non- or ex-smoker (A light-smoker is defined as someone using 10.0 nicotine units or less per day for at least 90 days prior to the first study drug administration. An ex smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration)
6. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by an investigator
7. Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the physical examination (including vital signs) and/or ECG, as determined by an investigator

   Healthy subjects (Phase 1a):
8. Male or female, aged at least 18 years but not older than 55 years
9. Body mass index (BMI) within 18.0 kg/m2 to 32.0 kg/m2, inclusive

   HBV-infected subjects (Phase 1b):
10. Male or female, aged at least 18 years but not older than 65 years
11. BMI within 18.0 kg/m2 to 35.0 kg/m2, inclusive
12. Serum HBsAg positive at screening and at least 6 months prior to screening
13. Serum HBeAg positive and HBV DNA ≥ 20,000 IU/mL, or serum HBeAg negative and HBV DNA ≥ 2,000 IU /mL at screening
14. ALT and AST <5 times the upper limit of normal (ULN) at screening and prior to the first study drug administration

Exclusion Criteria:

All subjects:

1. Female who is lactating at screening
2. Female who is pregnant according to the pregnancy test at screening or prior to the first study drug administration
3. History of significant hypersensitivity to clevudine or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
4. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease
5. Presence of clinically significant muscle disorders, myopathies or other forms of liver disease
6. Presence of clinically significant ECG abnormalities at the screening visit, as defined by medical judgment
7. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration
8. Any history of tuberculosis
9. Inclusion in a previous cohort for this clinical study
10. Intake of an Investigational Product (IP) in the 28 days prior to the first study drug administration
11. Active illicit drug use including, but not limited to, cocaine, heroin and methamphetamine (the use of cannabinoid is acceptable)
12. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration
13. Donation of 500 mL or more of blood in the 56 days prior to the first study drug administration

    Healthy subjects (Phase 1a):
14. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
15. Any clinically significant illness in the 28 days prior to the first study drug administration
16. Presence or history of clinically significant gastrointestinal, liver or kidney disease, or surgery that may affect drug bioavailability
17. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus tests
18. Use of any prescription drugs including amiodarone (with the exception of hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the participant as healthy

    HBV-infected subjects (Phase 1b):
19. Significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic)
20. Use of amiodarone in the 28 days prior to the first study drug administration
21. Presence or history of clinically significant gastrointestinal or kidney disease, or surgery that may affect drug bioavailability
22. Cirrhosis of the liver as determined by one of the following:

    * A score greater than F2 for liver fibrosis by FibroScan or FibroSure test within 6 months prior to screening or at the time of screening OR
    * A score greater than F2 on liver biopsy within 12 months prior to screening or at the time of screening
23. Medical history or known presence of hepatocellular carcinoma
24. Previous treatment for hepatitis B virus, including nucleoside therapy
25. Acute infection or any other clinically significant illness within 14 days of randomization
26. History of organ transplantation
27. Uncontrolled hypertension
28. Positive screening results to HIV Ag/Ab combo, hepatitis C virus or hepatitis D virus tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who experienced at least 1 treatment-emergent adverse event (TEAE) | Through study completion, an average of 1 year
The percentage of subjects who experienced at least one treatment emergent serious AE (SAE). | Through study completion, an average of 1 year
Percentage of subjects who experienced a treatment-emergent dose limiting toxicity (DLT) | Through study completion, an average of 1 year
Percentage of subjects who experienced at least one treatment emergent Grade 1, 2, 3, 4 or 5 laboratory abnormality | Through study completion, an average of 1 year
Percentage of subjects who discontinued study drug due to a TEAE | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of ATI-2173 and clevudine in Single Dose Healthy Volunteers | Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours
Food effect on Peak plasma concentration (Cmax) of ATI-2173 and clevudine in Single Dose Healthy Volunteers | Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours
Peak plasma concentration (Cmax) of ATI-2173 and clevudine in Multiple Dose Healthy Volunteers | Day 1 & Day 14: Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours. Day 14 only: post-dose at 48, 72, 144, 216, and 312 hours
Peak plasma concentration (Cmax) of ATI-2173 and clevudine in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Time of maximum observed plasma concentration (Tmax) of ATI-2173 and clevudine in Single Dose Healthy Volunteers | Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours
Food Effect on Time of maximum observed plasma concentration (Tmax) of ATI-2173 and clevudine in Single Dose Healthy Volunteers | Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours
Time of maximum observed plasma concentration (Tmax) of ATI-2173 and clevudine in Multiple Dose Healthy Volunteers | Day 1 & Day 14: Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours. Day 14 only: post-dose at 48, 72, 144, 216, and 312 hours
Time of maximum observed plasma concentration (Tmax) of ATI-2173 and clevudine in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Area under plasma concentration time curve (AUC) of ATI-2173 and clevudine in Single Dose Healthy Volunteers | Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours
Food Effect on Area under the concentration time curve (AUC0-t) from time 0 (dose administration) to the time of last quantifiable concentration (TLQC) of ATI-2173 and clevudine | Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours
Food Effect on Area under the concentration time curve (AUC0-inf) extrapolated to infinity, calculated as AUC0-t + CLQC/λZ, where CLQC is the measured concentration at time TLQC in ATI-2173 and clevudine | Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours
Area under the concentration time curve from time 0 (dose administration) to 24 hours (AUC0-24) in ATI-2173 and clevudine in Multiple Dose Healthy Volunteers | Day 1 & Day 14: Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours. Day 14 only: post-dose at 48, 72, 144, 216, and 312 hours
Area under the concentration time curve from time 0 (dose administration) to 24 hours (AUC0-24) in ATI-2173 and clevudine in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Terminal elimination half-life (t1/2) of ATI-2173 in plasma in Single Dose Healthy Volunteers | Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 20, 24, 36, 48, 72, 96, and 120 hours
Terminal elimination half-life (t1/2) of ATI-2173 in plasma in Multiple Dose Healthy Volunteers | Day 1 & Day 14: Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours. Day 14 only: post-dose at 48, 72, 144, 216, and 312 hours
Terminal elimination half-life (t1/2) of ATI-2173 in plasma in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Trough Peak plasma concentration (Ctrough) of ATI-2173 and clevudine in Multiple Dose Healthy Volunteers | Pre-dose on days 3, 5, 7, 10, and 13.
Trough Peak plasma concentration (Ctrough) of ATI-2173 and clevudine in Multiple Dose HBV Infected Patients | Pre-dose on days 3, 5, 7, 10, 14 and 21
Minimum observed plasma concentration (Cmin) of ATI-2173 and clevudine in a dosing interval in Multiple Dose Healthy Volunteers | Day 1 & Day 14: Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours. Day 14 only: post-dose at 48, 72, 144, 216, and 312 hours
Minimum observed plasma concentration (Cmin) of ATI-2173 and clevudine in a dosing interval in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Cumulative amount of drug excreted in urine over all time intervals (Ae) in Single Dose Healthy Volunteers | Pre-dose, post-dose at 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, and 96-120 hours
Cumulative amount of drug excreted in urine over all time intervals (Ae) in Multiple Dose Healthy Volunteers | Pre-dose on Day 1, post-dose on Days 1 & 14 at 0-4, 4-8, 8-12, 12-24 hours
Cumulative amount of drug excreted in urine over all time intervals (Ae) in Multiple Dose HBV Infected Patients | Pre-dose on Day 1, post-dose on Days 1 & 28 at 0-4, 4-8 and 8-24 hours
Apparent metabolic clearance (mCLr) of clevudine in urine in Single Dose Healthy Volunteers | Pre-dose, post-dose at 0-4, 4-8, 8-12, 12-24, 24-48, 48-72, 72-96, and 96-120 hours
Apparent metabolic clearance (mCLr) of clevudine in urine in Multiple Dose Healthy Volunteers | Pre-dose on Day 1, post-dose on Days 1 & 14 at 0-4, 4-8, 8-12, 12-24 hours
Apparent metabolic clearance (mCLr) of clevudine in urine in Multiple Dose HBV Infected Patients | Pre-dose on Day 1, post-dose on Days 1 & 28 at 0-4, 4-8 and 8-24 hours
Accumulation ratio of ATI-2173 and clevudine in plasma (RAC) evaluated by comparing Day 14 (Ph1a) Cmax to Day 1 Cmax in Multiple Dose Healthy Volunteers | Day 1 & Day 14: Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours. Day 14 only: post-dose at 48, 72, 144, 216, and 312 hours
Accumulation ratio of ATI-2173 and clevudine in plasma (RAC) evaluated by comparing Day 28 (Ph1b) Cmax to Day 1 Cmax in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Accumulation ratio of ATI-2173 and clevudine in plasma (RAC) evaluated by comparing Day 14 (Ph1a) AUCtau to Day 1 AUC0-24 in Multiple Dose Healthy Volunteers | Day 1 & Day 14: Pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours. Day 14 only: post-dose at 48, 72, 144, 216, and 312 hours
Accumulation ratio of ATI-2173 and clevudine in plasma (RAC) evaluated by comparing Day 28 (Ph1b) AUCtau to Day 1 AUC0-24 in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Resistance Mutations in Multiple Dose HBV Infected Patients | Day -1, Day 1, Day 7, Day 14, Day 21, Day 28, Day 31, Day 37, Day 55, Day 111, Day 195
  To assess the emergence of resistance mutations in HBV-infected subjects. The frequency of targeted mutations may be calculated in each subject.
Maximum observed HBV DNA change (reduction) from baseline through Day 28 (Emax) in Multiple Dose HBV Infected Patients | Screening, Day -1, 7, 14, 21, 28
Maximum observed HBV DNA change (reduction) from baseline through end of study (Emax) in Multiple Dose HBV Infected Patients | Screening, Day -1, 7, 14, 21, 28, 31, 37, 55, 111, and 195
Time (day) of maximum observed effect through Day 28 (TEmax) in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours
Time (day) of maximum observed effect through end of study (TEmax) in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours
Area under the effect concentration time curve from time 0 (first dose administration) to Day 28 that is above baseline (AUEC) in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours
Area under the effect concentration time curve from time 0 (first dose administration) to end of study (24 weeks post last dose) that is above baseline (AUEC) in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Area under the effect concentration time curve from time 0 (first dose administration) to Day 28 that is below baseline (AUEC) in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours
Area under the effect concentration time curve from time 0 (first dose administration) to end of study (24 weeks post last dose) that is below baseline (AUEC) in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
Area under the effect concentration time curve from time 0 (first dose administration) to Day 28 (AUEC) in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours
Area under the effect concentration time curve from time 0 (first dose administration) to end of study (24 weeks post last dose) (AUEC) in Multiple Dose HBV Infected Patients | Day 1: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours; Day 28: pre-dose, post-dose at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 144, 216 and 312 hours
ALT/AST Concentration versus Time in Multiple Dose HBV Infected Patients | Screening, Day -1, 1, 3, 7, 10, 14, 21, 28, 34, 37, 41, and 55

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Mayers, MD, Study Director — Antios Therapeutics, Inc
Locations (3):
- Altasciences, Montreal, Quebec, Canada
- Republican Clinical Hospital "Timofei Mosneaga" Arensia EM Unit, Chisinau, Republic of Moldova, Moldova
- Medical Center of Limited Liability Company "Harmoniya krasy" Department of Clinical Trials, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peek SF, Cote PJ, Jacob JR, Toshkov IA, Hornbuckle WE, Baldwin BH, Wells FV, Chu CK, Gerin JL, Tennant BC, Korba BE. Antiviral activity of clevudine [L-FMAU, (1-(2-fluoro-5-methyl-beta, L-arabinofuranosyl) uracil)] against woodchuck hepatitis virus replication and gene expression in chronically infected woodchucks (Marmota monax). Hepatology. 2001 Jan;33(1):254-66. doi: 10.1053/jhep.2001.20899. PMID 11124844
- [Background] Marcellin P, Mommeja-Marin H, Sacks SL, Lau GK, Sereni D, Bronowicki JP, Conway B, Trepo C, Blum MR, Yoo BC, Mondou E, Sorbel J, Snow A, Rousseau F, Lee HS. A phase II dose-escalating trial of clevudine in patients with chronic hepatitis B. Hepatology. 2004 Jul;40(1):140-8. doi: 10.1002/hep.20257. PMID 15239097
- [Background] Lee HS, Chung YH, Lee K, Byun KS, Paik SW, Han JY, Yoo K, Yoo HW, Lee JH, Yoo BC. A 12-week clevudine therapy showed potent and durable antiviral activity in HBeAg-positive chronic hepatitis B. Hepatology. 2006 May;43(5):982-8. doi: 10.1002/hep.21166. PMID 16628625
- [Background] Lim SG, Leung N, Hann HW, Lau GK, Trepo C, Mommeja-Marin H, Moxham C, Sorbel J, Snow A, Blum MR, Rousseau F, Marcellin P. Clinical trial: a phase II, randomized study evaluating the safety, pharmacokinetics and anti-viral activity of clevudine for 12 weeks in patients with chronic hepatitis B. Aliment Pharmacol Ther. 2008 Jun;27(12):1282-92. doi: 10.1111/j.1365-2036.2008.03686.x. Epub 2008 Mar 22. PMID 18363895
- [Background] Yoo BC, Kim JH, Chung YH, Lee KS, Paik SW, Ryu SH, Han BH, Han JY, Byun KS, Cho M, Lee HJ, Kim TH, Cho SH, Park JW, Um SH, Hwang SG, Kim YS, Lee YJ, Chon CY, Kim BI, Lee YS, Yang JM, Kim HC, Hwang JS, Choi SK, Kweon YO, Jeong SH, Lee MS, Choi JY, Kim DG, Kim YS, Lee HY, Yoo K, Yoo HW, Lee HS. Twenty-four-week clevudine therapy showed potent and sustained antiviral activity in HBeAg-positive chronic hepatitis B. Hepatology. 2007 May;45(5):1172-8. doi: 10.1002/hep.21629. PMID 17464992
- [Background] Yoo BC, Kim JH, Kim TH, Koh KC, Um SH, Kim YS, Lee KS, Han BH, Chon CY, Han JY, Ryu SH, Kim HC, Byun KS, Hwang SG, Kim BI, Cho M, Yoo K, Lee HJ, Hwang JS, Kim YS, Lee YS, Choi SK, Lee YJ, Yang JM, Park JW, Lee MS, Kim DG, Chung YH, Cho SH, Choi JY, Kweon YO, Lee HY, Jeong SH, Yoo HW, Lee HS. Clevudine is highly efficacious in hepatitis B e antigen-negative chronic hepatitis B with durable off-therapy viral suppression. Hepatology. 2007 Oct;46(4):1041-8. doi: 10.1002/hep.21800. PMID 17647293
- [Background] Fleischer RD, Lok AS. Myopathy and neuropathy associated with nucleos(t)ide analog therapy for hepatitis B. J Hepatol. 2009 Oct;51(4):787-91. doi: 10.1016/j.jhep.2009.06.011. Epub 2009 Jul 1. PMID 19665816
- [Background] Kim BK, Oh J, Kwon SY, Choe WH, Ko SY, Rhee KH, Seo TH, Lim SD, Lee CH. Clevudine myopathy in patients with chronic hepatitis B. J Hepatol. 2009 Oct;51(4):829-34. doi: 10.1016/j.jhep.2009.04.019. Epub 2009 May 28. PMID 19615776
- [Background] Seok JI, Lee DK, Lee CH, Park MS, Kim SY, Kim HS, Jo HY, Lee CH, Kim DS. Long-term therapy with clevudine for chronic hepatitis B can be associated with myopathy characterized by depletion of mitochondrial DNA. Hepatology. 2009 Jun;49(6):2080-6. doi: 10.1002/hep.22959. PMID 19333909
- [Background] Wang L, Sun R, Eriksson S. The kinetic effects on thymidine kinase 2 by enzyme-bound dTTP may explain the mitochondrial side effects of antiviral thymidine analogs. Antimicrob Agents Chemother. 2011 Jun;55(6):2552-8. doi: 10.1128/AAC.00109-11. Epub 2011 Mar 28. PMID 21444706
- [Background] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Background] PEGASYS® (peginterferon alfa-2a) Injection, for Subcutaneous Use. Initial U.S. Approval: 2002 Prescribing Information. https://www.gene.com/patients/medicines/pegasys
- [Background] Lok AS, Zoulim F, Dusheiko G, Ghany MG. Hepatitis B cure: From discovery to regulatory approval. Hepatology. 2017 Oct;66(4):1296-1313. doi: 10.1002/hep.29323. Epub 2017 Aug 1. PMID 28762522
- [Background] Terrault NA, Lok ASF, McMahon BJ, Chang KM, Hwang JP, Jonas MM, Brown RS Jr, Bzowej NH, Wong JB. Update on prevention, diagnosis, and treatment of chronic hepatitis B: AASLD 2018 hepatitis B guidance. Hepatology. 2018 Apr;67(4):1560-1599. doi: 10.1002/hep.29800. No abstract available. PMID 29405329
- [Background] VIREAD® (tenofovir disoproxil fumarate), Initial U.S. Approval 2001 Prescribing Information. https://www.gilead.com/science-and-medicine/- /media/files/pdfs/medicines/hiv/viread/viread_pi.pdf?la=en
- [Background] BARACLUDE® (entecavir), Initial U.S. Approval 2005 Prescribing Information. https://packageinserts.bms.com/pi/pi_baraclude.pdf
- [Derived] Squires KE, Ogilvie L, Jucov A, Anastasiy I, Ghicavii N, Huguet J, Melara R, Constantineau M, De La Rosa A, Mayers DL. A randomized phase 1b trial of the active site polymerase inhibitor nucleotide ATI-2173 in patients with chronic hepatitis B virus infection. J Viral Hepat. 2023 Jan;30(1):19-28. doi: 10.1111/jvh.13753. Epub 2022 Oct 22. PMID 36201354